CLINICAL TRIAL: NCT01241396
Title: An Observational Study of the Treatment of Multiple Myeloma in Routine Clinical Practice
Brief Title: A Study to Record in an Observational Manner the Treatment of Multiple Myeloma as it is Being Done in Every Day Practice Without Providing Any Investigational Drug or Prescribing Any Procedure
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017410
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; observational; survey; non-interventional; international; epidemiology; treatment; routine clinical practice; retrospective; prospective
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: Any MMY treatment Any line of treatment for MMY
  Interventions: Other: Any MMY treatment

INTERVENTIONS:
Other: Any MMY treatment — Any line of treatment for MMY

SUMMARY:
The primary objective of this observational study is to document and describe current treatment regimens and disease progression of patients with Multiple Myeloma (MMY). The aim of this registry is to provide accurate, descriptive information on the way Multiple Myeloma is treated in routine clinical practice. The registry will collect information related to the treatment received for Multiple Myeloma. About 3000 patients will take part in the study in about 28 countries. The registry will only collect information that is already in medical files regarding treatment. Patients will not be required to actively do anything in addition to what would be done without participating in this registry, nor will there be any procedures or interventions that are not already part of the current treatment.

DETAILED DESCRIPTION:
There is a lack of objective data relating to variation in treatment practices and resource utilisation for Multiple Myeloma (MMY) patients between countries. This void continues to hamper attempts to create meaningful health economic models for MMY treatment and impedes understanding of the MMY clinical arena. This non-interventional observational study is designed to address the problem by providing a definitive picture of routine treatment and resource utilisation practices for MMY patients at any stage of treatment, independent of drug(s) used and treatment line across the different countries taking part. A non-interventional study design has been selected to facilitate data collection about routine clinical practice. This study seeks to obtain an appropriate subset of the true population of patients with MMY throughout Europe Middle East and Africa. Many concerns exist when attempting to develop an unbiased study sample, including biases regarding the selection of patients to be enrolled. Therefore, a multi-staged site and patient selection model will be used to reduce biases associated with patient and site selection. The study seeks to enroll at least 3,000 patients. It will deliver a description of everyday treatment practice of MMY. Additional retrospective medical reviews will also be performed to collect information regarding disease history. The primary objective of the study is to document and describe current treatment regimens and disease progression of patients with MMY. Secondary objectives of the study involve understanding the MMY patient population and its generalisability to all treated MMY patients. Additional goals of the study are to document and compare: (a) utilisation of current treatment regimens for MMY; (b) quality of life and health economic parameters associated with MMY treatment regimens; (c) the safety profile of current treatment regimens for MMY and the impact on resource utilisation; (d) the effectiveness of current treatment regimens for MMY. The study will collect prospective data on efficacy, outcomes, health economic and safety parameters for all patients whenever available. The resulting database will allow future health economic, pharmaco-epidemiological, and outcomes research, and provide important data from the clinical arena. At least 3000 patients will be recruited to this study. As this is an observational study, the decision of patients to take part in this study will not have any impact on the care they are receiving. All treatment decisions will be made at the discretion of the participating physicians. Only data available from routine clinical practice will be collected. There are two phases of data collection in this study: (a) at baseline, the patient's historical treatment and resource utilisation data, where possible stretching back to diagnosis, will be recorded via electronic data capture; (b) following the baseline visit, the patient will enter a prospective data collection phase where data will be collected at least every three months. At each data collection point, all changes since the previous data collection point will be collected. Prospective data collection will continue until the study is complete or the patient is withdrawn from the study. Data will continue to be captured until three years after the last patient is recruited to the study. Interim analyses will be conducted at least annually to update the current data. To monitor the safety profile of MMY treatment related to a Johnson and Johnson product, any unwanted effects that occur during the MMY treatment will be recorded Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

- Requires commencement of a new line of treatment for MMY at any stage, regardless of type of therapy selected.

Exclusion Criteria:

* Patients currently participating in another investigational study or clinical trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will focus on enrolling consecutively, patients who are initiating any new line of therapy for Multiple Myeloma, regardless of the line of treatment. Because this is a non-interventional study, intended to provide a picture of routine clinical practice, no guidance will be given on any aspect of treatment, patient clinical management or treatment dose selection.
Sampling Method: Probability Sample
Enrollment: 2396 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Description of current treatment regimens for MMY. | Every 3 months from baseline to 3 years after last patient recruited

SECONDARY OUTCOMES:
Utilisation of current treatment regimens for MMY | Every 3 months from baseline to 3 years after last patient recruited
Quality of life and health economic parameters associated with MMY treatment regimens | Every 3 months from baseline to 3 years after last patient recruited
Safety profile of current treatment regimens for MMY | Every 3 months from baseline to 3 years after last patient recruited
The effectiveness of current treatment regimens for MMY | Every 3 months from baseline to 3 years after last patient recruited

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (159):
- Algeria (5):
  - Algiers
  - Constantine
  - Oran
  - Sétif
  - Tizi Ouzou
- Austria (2):
  - Graz
  - Innsbruck
- Zagreb, Croatia
- Denmark (2):
  - Holstebro
  - Odense
- Estonia (2):
  - Tallinn
  - Tartu
- France (14):
  - Avignon
  - Blois
  - Bordeaux
  - Brest
  - Clermont-Ferrand
  - Le Mans
  - Montpellier
  - Nantes
  - Nîmes
  - Perpignan
  - Pontoise
  - Rennes
  - Saint-Brieuc
  - Troyes
- Germany (36):
  - Amberg
  - Aschaffenburg
  - Augsburg
  - Bad Soden
  - Bamberg
  - Berlin
  - Bielefeld
  - Bonn
  - Borken
  - Bottrop
  - Bremerhaven
  - Coburg
  - Dresden
  - Goslar
  - Hamburg
  - Hamm
  - Hanover
  - Hildesheim
  - Hof
  - Kaiserslautern
  - Lübeck
  - Mainz
  - Mayen
  - Mutlangen
  - München
  - Naunhof
  - Neunkirchen
  - Nuremberg
  - Olpe
  - Ostfildern
  - Rostock
  - Rotenburg (Wümme)
  - Saarbrÿcken
  - Stuttgart
  - Weiden
  - Würzburg
- Greece (3):
  - Athens
  - Larissa
  - Thessalonikis
- Hungary (5):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
  - Szombathely
- Israel (4):
  - Haifa
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
- Riga, Latvia
- Lithuania (2):
  - Klaipėda
  - Vilnius
- Skopje, North Macedonia
- Poland (17):
  - Bialystok
  - Brzozów
  - Bytom
  - Chorzów
  - Gdansk
  - Gorzów Wielkopolski
  - Katowice
  - Legnica
  - Lublin
  - Opole
  - Poznan
  - Rzeszów
  - Słupsk
  - Warsaw
  - Warszawa Poland
  - Wroclaw
  - Zamość
- Portugal (2):
  - Ponta Delgada
  - Porto
- Russia (12):
  - Kolomna
  - Krasnodar
  - Krasnogorsk
  - Moscow
  - Podolsk
  - Saint Petersburg
  - Samara
  - Saransk
  - Tula
  - Ulyanovsk
  - Volgograd
  - Vologda
- Ljubljana, Slovenia
- South Africa (4):
  - Bloemfontein
  - Cape Town
  - Durban
  - Johannesburg
- Spain (18):
  - Alicante
  - Barcelona
  - Cadiz
  - Cáceres
  - Ciudad Real
  - Donostia / San Sebastian
  - Guadalajara
  - Jaén
  - León
  - Madrid
  - Marbella
  - Murcia
  - Palma de Mallorca
  - Salamanca
  - Seville
  - Talavera de La Reina, Toledo
  - Tarragona
  - Zaragoza
- Turkey (Türkiye) (8):
  - Adana
  - Ankara
  - Antalya
  - Bursa
  - Istanbul
  - Izmir
  - Kayseri
  - Samsun
- Ukraine (19):
  - Cherkassy
  - Dnipro
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kherson
  - Khmelnitskiy
  - Kiev
  - Lutsk
  - Lviv
  - Mykolayiv
  - Odesa
  - Poltava
  - Simferopol
  - Ternopil
  - Uzhhorod
  - Vinnitsa
  - Zaporizhzhya
  - Zhytomyr